CLINICAL TRIAL: NCT05675826
Title: The Impact of Donor COVID-19 Infection Status on the Recipient in Allogeneic Hematopoietic Stem Cell Transplantation.
Brief Title: The Impact of Donor COVID-19 Infection Status on the Recipient in Allo-HSCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chen Suning (Other)
Responsible Party: Sponsor-Investigator, Chen Suning, Physician, The First Affiliated Hospital of Soochow University
Organization: The First Affiliated Hospital of Soochow University (Other)
Other Study IDs: COVID19-HSCT-1
Record Dates: First submitted 2023-01-04; First posted 2023-01-09 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: COVID-19; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Donor infected with covid19: This includes donors who have been infected or are infected with COVID19 at the time of hematopoietic stem cell collection.
- Donor not infected with covid: Including donors not yet infected with COVID19 at the time of hematopoietic stem cell collection.

SUMMARY:
This study was conducted to observe whether COVID-19 can be transmitted through stem cell transplantation and whether COVID-19-positive donors have an effect on early hematopoietic reconstitution and immune reconstitution in the recipients.

DETAILED DESCRIPTION:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) induced COVID-19 infections are showing an explosive increase in China starting in late 2022. SARS-CoV-2 infections are characterized by an initial viral replication followed by an inflammatory phase with lymphocyte depletion in severe patients.

Past studies have shown that SARS-CoV -2 is detectable in the blood of 8%-15% of patients and that viremia occurs in the first 2-3 days after the onset of symptoms. EBMT, WMDA and other organizations have suggested that COVID-19 positive donors must be excluded or delayed from donation for safety reasons.

However, there have not been any reports of transmission from donor to recipient in blood product transfusion or cell therapy. In the only reported cases of allogeneic HSCT from SARS-CoV-2 positive donors, there was also no evidence of recipient infection from the graft.

In the current situation where the vast majority of people are infected with COVID-19 in the short term, many patients, such as those with leukemia, are in urgent need of transplantation due to the aggressive， hard-to-control，underlying disease. The investigators established this observational clinical trial to investigate whether COVID-19 is transmitted through stem cells and whether COVID-19 positive donors have an impact on early hematopoietic reconstitution and immune reconstitution in recipients.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 16 and 65 years old.
2. History of hematological malignancies (acute leukemias, myelodysplastic syndromes, myeloproliferative neoplasms, lymphomas, myeloma).
3. Allogeneic hematopoietic stem cell transplantation perform during the COVID19 pandemic.

Exclusion Criteria:

Hematological diseases, other than hematological malignancies.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population wil be patients who underwent allogeneic HSCT during the COVID19 epidemic.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-12-26 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Hematopoietic reconstitution | 1 month after enrollment of the last case
  To compare the differences in the time of hematopoietic reconstitution between the two groups after transplantation.

SECONDARY OUTCOMES:
Infection of COVID19 | 1 month after enrollment of the last case
  To compare the rate of early COVID19 infection between the two groups as well as the rate of severe disease.
Acute graft-versus-host disease | 100 days after enrollment of the last case
  To compare the incidence and extent of aGVHD between the two groups.
COVID19 related mortality | 100 days after enrollment of the last case
  The percentage of HM patients with COVID-19 who died.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China